CLINICAL TRIAL: NCT05071820
Title: Validation of a Microlearning Approach to a Diabetes Prevention Program
Brief Title: Microlearning Application for Diabetes Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators decided to halt the study early because the company delivering the microlearning platform was incorporated into another company.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sandra Anping Tsai, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61279
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: PreDiabetes; Elevated Blood Sugar
MeSH Terms: conditions — Prediabetic State; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application program (Experimental)
  Interventions: Other: Health U mobile application
- Traditional program (Active Comparator)
  Interventions: Other: National Diabetes Prevention Program

INTERVENTIONS:
Other: Health U mobile application — Health U mobile application delivers daily microlearning modules and the health coach interactions within the Health U application
  Arms: Mobile application program
Other: National Diabetes Prevention Program — CDC recognized National DPP that follows a set curriculum with modules delivered over 12 months
  Arms: Traditional program

SUMMARY:
The purpose of this study is to test the effectiveness of a mobile application diabetes prevention program delivered with microlearning and microcoaching.

DETAILED DESCRIPTION:
Patients with prediabetes who are interested in joining a diabetes prevention program will be randomized to either the mobile application diabetes prevention program or the traditional diabetes prevention program, which is delivered as a mixed program of in-person and virtual sessions.

Study participants in the mobile application version will download the Health U app from the Apple application store. The user will complete the daily microlearning modules and the health coach interactions within the Health U application. The 12-month diabetes prevention program will follow the widely clinically-validated CDC Get Active to Prevent T2 curriculum.

For participants participating in the in-person version, they will complete the diabetes prevention program, which meets in-person and virtually approximately once every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years old
* high risk for type 2 diabetes (history of gestational diabetes, A1c 5.7-6.4)

Exclusion Criteria:

* pregnant
* non-English speaker
* not comfortable using a mobile application

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Percent weight lost at 12 months from baseline weight | 12 months

SECONDARY OUTCOMES:
change in hemoglobin A1c | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Tsai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No